CLINICAL TRIAL: NCT01441115
Title: Phase I Trial of ECI301 in Combination With Radiation in Patients With Advanced or Metastatic Cancer
Brief Title: ECI301 and Radiation for Advanced or Metastatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A trial using ECI301 & radiation was initiated in Japan in 2012. This tested the primary endpoint in a duplicate trial, thus the study was closed.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Deborah Citrin, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110248; 11-C-0248
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Results first posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-11

CONDITIONS: Cancer; Neoplasm Metastasis; Radiation Oncology; Neoplasm; Metastasis
Keywords: Metastasis; Cancer; Radiation Therapy; Locally Advanced; Palliation; Metastatic Cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ECI301 Dose level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer (Experimental): ECI301 Dose level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer
  Interventions: Procedure: Radiation Therapy; Drug: ECI301

INTERVENTIONS:
Procedure: Radiation Therapy
Drug: ECI301

SUMMARY:
Background:

- ECI301 is a drug that may help make cancer cells more visible to the immune system after radiation. The drug may also help the immune system destroy the cancer at sites that have not received radiation therapy. Researchers want to study ECI301 in people with advanced cancer or cancer that has spread in the body (metastatic).

Objectives:

- To test ECI301 with radiation therapy for advanced or metastatic cancer.

Eligibility:

- People at least 18 years of age with either metastatic or advanced cancer that may benefit from radiation therapy.

Design:

* Participants will be screened with a medical history and physical exam. They will also have blood and urine tests, and imaging studies.
* All participants will have radiation therapy 5 days a week for 2 weeks.
* They will have different doses of ECI301 to test its safety and effectiveness. ECI301 will be given in a vein during the second week of radiation therapy. Frequent blood tests and imaging studies will monitor the treatment.
* After participants have ECI301, tumor samples may be taken from the site that had radiation and another site that did not have radiation.
* Follow-up visits will include blood tests and imaging studies.

DETAILED DESCRIPTION:
Background:

* Patients with metastatic or locally advanced cancer frequently require palliative radiotherapy to relieve symptoms; however, progression of disease is frequent in patients with extended survival
* Radiation results in tumor cell death which can result in increased dendritic cell activation and trafficking
* ECI301 is a derivative of Macrophage Inflammatory Protein-1 alpha, a 70 amino acid chemokine that is a ligand for C-C chemokine receptor type 1 (CCR1) and C-C chemokine receptor type 5 (CCR5), the chemokine receptors of immature dendritic cells.
* ECI301 has been shown to enhance the effect of radiotherapy in animal models.

Objectives:

* The primary objective is to determine the maximum tolerated dose (MTD) of ECI301 delivered in combination with 30 Gray (Gy) of external beam radiation to patients with metastatic or locally advanced cancer.
* The secondary objectives are:

  * To describe the safety and tolerability of ECI301 delivered in combination with 30 Gy of external beam radiation to patients with metastatic or locally advanced cancer
  * To evaluate the humoral and cellular immune responses by:

    * Measurement of circulating precursor dendritic cells before and after the completion of ECI301
    * Measurement of circulating MIP-alpha before and after the completion of ECI301
    * Assessment of T-lymphocyte quantitative and qualitative changes by flow cytometry and assays for interferon (IFN-gamma) production
  * To define pharmacologic parameters following the intravenous dose of ECI301
  * To determine if neutralizing anti-EC301 antibodies occur after treatment
  * To describe the response at the radiated site and distant sites after radiation in combination with ECI301

Eligibility:

* Age >18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <2.
* Life expectancy of greater than 3 months
* Histologically confirmed metastatic or locally advanced cancer for which radiotherapeutic management would be appropriate
* No recent history of myocardial infarction or unstable angina

Design:

* This is a Phase I trial to determine the maximum tolerated dose of ECI301 in combination with external beam radiation therapy in patients with locally advanced or metastatic solid tumors.
* Patients will be treated with radiation therapy in a standard manner with ECI301 given daily during radiation. The dose of ECI301 will be escalated over the course of the trial to determine the maximum tolerated dose (MTD of daily ECI301 in combination with radiotherapy.
* We anticipate that accrual to this trial of 30 patients will take approximately 2 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

2.1.1.1 Age greater than or equal to18 years.

2.1.1.2 Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.

2.1.1.3 Life expectancy of greater than 3 months

2.1.1.4 Histologically confirmed cancer

2.1.1.5 Extracranial metastatic cancer or locally advanced cancer for which palliative radiotherapeutic management would be appropriate (no more than two sites will be treated on this trial)

2.1.1.6 Patients must have measurable or evaluable disease at the site(s) requiring radiation

2.1.1.7 Adequate marrow and organ function defined as

* absolute neutrophil count (ANC) > 1.5 times 10(9)/L,
* platelet count > 100 times 10(9),
* hemoglobin >9 g/L.
* creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal
* serum bilirubin <1.5 times upper limit reference range (ULRR),
* alanine aminotransferase (ALT), aspartate aminotransferase (AST), or

alkaline phosphatase (ALP) <2.5 times the ULRR (<5 times the ULRR in the presence

of liver metastases)

2.1.1.8 Female patients of childbearing potential must either be surgically sterile to prevent pregnancy, be at least 1-year post-menopausal, or have had no menses for 12 months, or agree to use reliable methods of contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, copper banded intrauterine device, tubal ligation or abstinence) from time of screening until 4 weeks after discontinuing study treatment. It is not known whether ECI301 has the capacity to induce hepatic enzymes so hormonal contraceptives should be combined with a barrier method of contraception.

2.1.1.9 Male patients must agree to use barrier contraception (i.e. condoms) and refrain from donating sperm from the start of dosing until 16 weeks after discontinuing study treatment. If male patients wish to father children, they should be advised to arrange for freezing of sperm prior to the start of study treatment.

EXCLUSION CRITERIA:

2.1.2.1 Pregnant or lactating females

2.1.2.2 Contraindications to radiotherapy (i.e. prior radiotherapy to the intended treatment site)

2.1.2.3 Untreated or previously treated but progressive intracranial metastases (Patients with previously treated intracranial metastases should have no clinical evidence of progression and be at least 4 weeks from therapy for intracranial metastases)

2.1.2.4 Need for emergent radiotherapy (defined as need for radiotherapy within 24 hours of consultation at the judgment of the treating radiation oncologist)

2.1.2.5 Active treatment with immunosuppressive therapy and subjects taking systemic corticosteroid therapy for any reason including replacement therapy for hypoadrenalism

2.1.2.6 Chemotherapy, radiation therapy, Tamoxifen or investigational therapy during the 4 weeks prior to initiation of protocol therapy

2.1.2.7 History of rheumatoid arthritis, systemic lupus erythematosus, Sjogren's disease, sarcoidosis, vasculitis, polymyositis, temporal arteritis or any other autoimmune disease

2.1.2.8 History of organ transplant

2.1.2.9 Human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C positivity

2.1.2.10 Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

2.1.2.11 Use of excluded immune modulating medications within 4 weeks prior to protocol therapy, or requirement for concurrent use.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-09-06 (Actual); Primary Completion 2013-04-24 (Actual); Study Completion 2013-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Citrin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman EJ. Immune modulation by ionizing radiation and its implications for cancer immunotherapy. Curr Pharm Des. 2002;8(19):1765-80. doi: 10.2174/1381612023394089. PMID 12171547
- [Background] Sharp HJ, Wansley EK, Garnett CT, Chakraborty M, Camphausen K, Schlom J, Hodge JW. Synergistic antitumor activity of immune strategies combined with radiation. Front Biosci. 2007 Sep 1;12:4900-10. doi: 10.2741/2436. PMID 17569618
- [Background] Maurer M, von Stebut E. Macrophage inflammatory protein-1. Int J Biochem Cell Biol. 2004 Oct;36(10):1882-6. doi: 10.1016/j.biocel.2003.10.019. PMID 15203102

RESULTS

PARTICIPANT FLOW:
Groups:
- ECI301 Dose Level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer: ECI301 Dose level 1 - 25 ug/kg and radiation therapy for advanced or metastatic cancer.
Period: Overall Study
Arm/Group | ECI301 Dose Level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer
Started | 2
Completed | 1
Not Completed | 1
Not completed — Taken off study - Principal Investigator discretion | 1

BASELINE CHARACTERISTICS:
Arm/Group | ECI301 Dose Level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of ECI301 Delivered in Combination With 30 Gray (Gy) External Beam Radiation to Participants With Metastatic or Locally Advanced Cancer
Description: MTD is defined as the highest dose level at which no more than 1 of 6 participants experience dose-limiting toxicity (DLT) during treatment or the first three weeks after treatment, and the dose below that at which at least 2 (of ≤6) participants have DLT as a result of the drug. Examples of DLT is any grade 3 or greater non-hematologic toxicity, ang grade 3 neutropenia or thrombocytopenia, any grade 4 anemia, and toxicity requiring a cumulative radiation treatment delay of 4 or more days.
Time Frame: During treatment or the first three weeks after treatment
Population: This MTD was not found because the trial was terminated early. A trial using ECI301 & radiation was initiated in Japan in 2012. This tested the primary endpoint in a duplicate trial, thus the study was closed. In addition, as specified in the protocol, the number of participants required to complete this trial involves 5 cohorts of 3 to 6 participants.
Arm/Group | ECI301 Dose Level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Adverse Events Unrelated, Unlikely, and Possibly Related to ECI301 Delivered in Combination With 30 Gray (Gy) of External Beam Radiation to Participants With Metastatic or Locally Advanced Cancer
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0) and the Radiation Therapy Oncology Group (RTOG) criteria.
Time Frame: Date treatment consent signed to date off study, and up to 30 days following the last dose of study drug, approximately 5 months and 25 days.
Population: 1/2 participants were analyzed because one participant was taken off study per Principal Investigator discretion and did not receive drug.
Measure: Number; unit: Adverse events
Groups:
- Unrelated; Unlikely Related; Possibly Related: ECI301 Dose level 1 - 25 ug/kg and radiation therapy for advanced or metastatic cancer.
Arm/Group | Unrelated | Unlikely Related | Possibly Related
Number analyzed (Participants) | 1 | 1 | 1
Adverse events
  Alanine aminotransferase increased | 0 | 1 | 0
  Anemia | 4 | 0 | 0
  Aspartate aminotransferase increased | 0 | 1 | 0
  Edema limbs | 1 | 0 | 0
  Erythema multiforme | 0 | 0 | 1
  Gastritis | 0 | 1 | 0
  Headache | 1 | 0 | 0
  Hyperkalemia | 0 | 1 | 0
  Lymphocyte count decreased | 1 | 0 | 0
  Pain in extremity | 1 | 0 | 0
  Urinary tract infection | 0 | 0 | 1

3. Secondary Outcome: Humoral and Cellular Immune Responses
Description: Measurement of circulating precursor dendritic cells, circulating macrophage inflammatory protein-1 alpha (MIP-α), and assessment of T-lymphocytes will be measured by flow cytometry and assays for type II interferon (IFNγ) production.
Time Frame: Before and after completion of ECI301
Population: This outcome measure was not done because the trial was terminated early. A trial using ECI301 & radiation was initiated in Japan in 2012. This tested the primary endpoint in a duplicate trial, thus the study was closed. In addition, as specified in the protocol, the number of participants required to complete this trial involves 5 cohorts of 3 to 6 participants.
Arm/Group | ECI301 Dose Level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer
Number analyzed (Participants) | 0

4. Secondary Outcome: Pharmacologic Parameters Following the Intravenous Dose of ECI301
Description: Pharmacologic parameters will be derived using non-compartmental analysis.
Time Frame: Following the intravenous dose of ECI301
Population: as for outcome 3
Arm/Group | ECI301 Dose Level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Response at the Radiated Site and Distant Site After Radiation in Combination With ECI301
Description: Response will be measured by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progression. Stable disease is neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ECI301 Dose Level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer
Number analyzed (Participants) | 1
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 1
  Progressive Disease | 0

6. Other Pre Specified Outcome: Here is the Number of Participants With Non-Serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ECI301 Dose Level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer
Number analyzed (Participants) | 1
Participants | 1

7. Other Pre Specified Outcome: Number of Participants With a Dose-Limiting Toxicity (DLT)
Description: Examples of DLT is any grade 3 or greater non-hematologic toxicity, any grade 3 neutropenia or thrombocytopenia, any grade 4 anemia; nausea, vomiting, diarrhea, tumor pain, or pre-existing hyponatremia, dyselectrolytemia, or orthostatic hypotension that has been optimally treated with anti-emetics, anti-diarrheal, analgesics, or hydration and which persists for over 48 hours despite maximal medical therapy, and toxicity requiring a cumulative radiation treatment delay of 4 or more days.
Time Frame: During treatment or the first three weeks after treatment
Population: 1/2 participants was analyzed because one participant was taken off study per Principal Investigator discretion and did not receive drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ECI301 Dose Level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, and up to 30 days following the last dose of study drug, approximately 5 months and 25 days.
Description: 1/2 participants were analyzed because one participant was taken off study per Principal Investigator discretion and did not receive drug.
Groups:
- ECI301 Dose Level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer: ECI301 Dose level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer
  Radiation Therapy
  ECI301
Arm/Group | ECI301 Dose Level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECI301 Dose Level 1 - 25 ug/kg and Radiation for Advanced or Metastatic Cancer (N=1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2011-11-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT01441115/Prot_SAP_000.pdf
  • Informed Consent Form (2011-11-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT01441115/ICF_001.pdf